CLINICAL TRIAL: NCT03467230
Title: Performance Assessment of the PMD-200 in Subjects Requiring Surgery Under General Anesthesia
Brief Title: Performance Assessment of the PMD-200 Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Borzoo Farhang, Assistant Professor of Anesthesiology, University of Vermont
Other Study IDs: 18-0302
Record Dates: First submitted 2018-02-27; First posted 2018-03-15 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Pain; Opioid Use; Intraoperative Complications
MeSH Terms: conditions — Pain; Intraoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NoL Index: All patients will be monitored by PMD-200 device
  Interventions: Device: NoL Index

INTERVENTIONS:
Device: NoL Index — Use of the PMD-200 in an observational study

SUMMARY:
A novel measure of nociception is the nociception level (NoL) index. The NoL index ranges from 0 to 100 and is based on a combination of nociception-related physiologic variables, which estimates the nociceptive/antinociceptive state.

The purpose of this project is to conduct an observational study of the PMD-200 noninvasive monitor (Medasense Biometrics Ltd., Ramat Gan, Israel), As this is an observational study, this monitor will not be used for clinical decision making, and the point of the study is to assess what happens with the NoL index during routine care. After thorough discussion with patients and written informed consent is provided in the pre-operative unit, patients will be transferred to the operating room. Patients will be connected to a vital sign monitor and any other medical equipment needed for the surgical procedure, as required by the standard of practice. The PMD-200 finger probe will be connected to the left hand middle finger (or right). The PMD-200 will be activated after the induction of general anesthesia. A calibration period of 1-2 minutes will be performed. At the conclusion of the surgical procedure, the PMD200 will be disconnected from the patient.

All the phases of anesthetic care are performed at the discretion of the anesthesiologist, but the time of administration of analgesics, muscle relaxants and other medications during anesthetic care will be recorded. The investigators will also record the time point of intubation (placement of breathing tube), extubation (removal of breathing tube), skin incision and any other significant surgical stimulation or noxious stimulation during the procedure. The investigators will be comparing NOL values prior to and following noxious stimuli, administration of analgesic agents and during non-noxious periods.

DETAILED DESCRIPTION:
The primary efficacy objective of this study is to demonstrate that the NOL Index of the PMD-200 monitor (Medasense Biometrics Ltd., Ramat Gan, Israel) is correlated with the responses to noxious stimuli and analgesic administration during the surgical procedure (prior and following a stimuli or titration), and the secondary efficacy objective of the study is to determine whether the NOL values can be correlated to other nociception predictors (e.g., increase in heart rate or blood pressure) following a noxious stimuli. The primary safety objective of this study is to assess the rate of any adverse reaction related to the study device. This device will not be used to make any clinical decision.

General anesthesia is the combination of various components including lack of movement, hypnosis, amnesia, control of autonomic responses, and attenuation of the response to noxious stimulation. Some anesthetic components, such as muscle relaxation and absence of movement are easy to assess with a twitch monitor. Similarly, hypnotic state can be estimated using processed electroencephalographic signals, but the anesthetic component that remains the most challenging to assess is the nociceptive/antinociceptive state. Typically, intraoperative nociception is estimated from autonomic responses (such as change in blood pressure and heart rate) and clinical signs such as tearing and sweating, but these variables can be very unreliable in predicting pain such as in patients who take beta blockers for treatment of high blood pressure whose heart rate may not increase in response to pain, patients with significant bleeding during surgery whose blood pressure may not increase in response to pain, etc. Effective antinociception is an important component of balanced anesthesia and appears to enhance postoperative outcomes. The most obvious potential consequence of insufficient intraoperative antinociceptive treatment is excessive postoperative pain, but inadequate treatment may also promote inflammatory, hormonal, and immunologic imbalances.

A novel measure of nociception is the nociception level (NoL) index. The NoL index ranges from 0 to 100 and is based on a nonlinear combination of nociception-related physiologic variables, specifically heart rate (HR), heart rate variability at the 0.15- to 0.4-Hz band power, photoplethysmograph wave amplitude (PPGA), skin conductance level, number of skin conductance fluctuations, and their time derivatives. The NoL index estimates the nociceptive/antinociceptive state from these components measures using random forest regression. Previous experimental work on a small number of patients showed that the NoL index is superior to each individual component and to a linear combination of the components. However, it remains unknown whether the NoL index accurately quantifies patients' intraoperative responses to noxious stimuli of varying intensities. The investigators therefore wish to evaluate the ability of the NoL index to discriminate noxious from nonnoxious stimuli, respond to analgesic administration, and progressively increase in response to increasing intensity of noxious stimulation.

In this observational study, The investigators attempt to learn the proper use of the PMD-200 and assess safety and efficacy of this device as mentioned above; however, no clinical decision will be based on the NoL index obtained.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Requiring laparoscopic gastrointestinal or laparoscopic hysterectomy under general anesthesia (without regional anesthesia)
* Patient provides informed consent

Exclusion Criteria:

* History of severe cardiac arrhythmias within the last 12 months
* Chronic pain conditions or analgesic usage (>1 month of large doses of opioids: more than 30mg oral equivalent of morphine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients ASA I-III scheduled for general anesthesia for laparoscopic GI or GU procedures.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy objective: Correlation of NoL Index with noxious stimulation/analgesic use | Intraoperatively
  To demonstrate that the NOL Index of the PMD-200 monitor (Medasense Biometrics Ltd., Ramat Gan, Israel) is correlated with the responses to noxious stimuli and analgesic administration during the surgical procedure (prior and following a stimuli or titration). Specifically, the investigators will assess the % change from baseline-steady state NoL Index value with the NoL Index value during surgical stimulation (increased noxious stimulation) as well as the NoL Index value after administration of analgesics (decreased noxious stimulation).

SECONDARY OUTCOMES:
the secondary efficacy objective: Correlation of NoL Index with changes in heart rate | Intraoperatively
  To determine whether the NOL values can be correlated to other nociception predictors (increase in heart rate) following a noxious stimuli.
the secondary efficacy objective: Correlation of NoL Index with blood pressure | Intraoperatively
  To determine whether the NOL values can be correlated to other nociception predictors (increase in blood pressure) following a noxious stimuli.
Safety objective: Any adverse reaction related to device | Intraoperatively
  To assess the rate of any adverse reaction related to the study device, any skin irritation or other unforeseen adverse reactions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Borzoo Farhang, DO, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ben-Israel N, Kliger M, Zuckerman G, Katz Y, Edry R. Monitoring the nociception level: a multi-parameter approach. J Clin Monit Comput. 2013 Dec;27(6):659-68. doi: 10.1007/s10877-013-9487-9. Epub 2013 Jul 9. PMID 23835792
- [Background] Martini CH, Boon M, Broens SJ, Hekkelman EF, Oudhoff LA, Buddeke AW, Dahan A. Ability of the nociception level, a multiparameter composite of autonomic signals, to detect noxious stimuli during propofol-remifentanil anesthesia. Anesthesiology. 2015 Sep;123(3):524-34. doi: 10.1097/ALN.0000000000000757. PMID 26154185
- [Background] Edry R, Recea V, Dikust Y, Sessler DI. Preliminary Intraoperative Validation of the Nociception Level Index: A Noninvasive Nociception Monitor. Anesthesiology. 2016 Jul;125(1):193-203. doi: 10.1097/ALN.0000000000001130. PMID 27171828
- [Background] Rantanen M, Yli-Hankala A, van Gils M, Ypparila-Wolters H, Takala P, Huiku M, Kymalainen M, Seitsonen E, Korhonen I. Novel multiparameter approach for measurement of nociception at skin incision during general anaesthesia. Br J Anaesth. 2006 Mar;96(3):367-76. doi: 10.1093/bja/ael005. Epub 2006 Jan 23. PMID 16431883
- [Background] Loeser JD, Treede RD. The Kyoto protocol of IASP Basic Pain Terminology. Pain. 2008 Jul 31;137(3):473-477. doi: 10.1016/j.pain.2008.04.025. Epub 2008 Jun 25. No abstract available. PMID 18583048
- [Background] Le Guen M, Liu N, Bourgeois E, Chazot T, Sessler DI, Rouby JJ, Fischler M. Automated sedation outperforms manual administration of propofol and remifentanil in critically ill patients with deep sedation: a randomized phase II trial. Intensive Care Med. 2013 Mar;39(3):454-62. doi: 10.1007/s00134-012-2762-2. Epub 2012 Dec 6. PMID 23223772
- [Background] Salo M. Effects of anaesthesia and surgery on the immune response. Acta Anaesthesiol Scand. 1992 Apr;36(3):201-20. doi: 10.1111/j.1399-6576.1992.tb03452.x. PMID 1574967
- [Background] Libby P. Inflammation in atherosclerosis. Nature. 2002 Dec 19-26;420(6917):868-74. doi: 10.1038/nature01323. PMID 12490960
- [Background] Vallejo R, Hord ED, Barna SA, Santiago-Palma J, Ahmed S. Perioperative immunosuppression in cancer patients. J Environ Pathol Toxicol Oncol. 2003;22(2):139-46. doi: 10.1615/jenvpathtoxoncol.v22.i2.70. PMID 14533877
- [Background] Tsuchiya Y, Sawada S, Yoshioka I, Ohashi Y, Matsuo M, Harimaya Y, Tsukada K, Saiki I. Increased surgical stress promotes tumor metastasis. Surgery. 2003 May;133(5):547-55. doi: 10.1067/msy.2003.141. PMID 12773983
- [Background] Page GG, Ben-Eliyahu S. The immune-suppressive nature of pain. Semin Oncol Nurs. 1997 Feb;13(1):10-5. doi: 10.1016/s0749-2081(97)80044-7. PMID 9048431
- [Background] Crozier TA, Muller JE, Quittkat D, Sydow M, Wuttke W, Kettler D. Effect of anaesthesia on the cytokine responses to abdominal surgery. Br J Anaesth. 1994 Mar;72(3):280-5. doi: 10.1093/bja/72.3.280. PMID 8130044
- [Background] Corsi M, Mariconti P, Calvillo L, Falchi M, Tiengo M, Ferrero ME. Influence of inhalational, neuroleptic and local anaesthesia on lymphocyte subset distribution. Int J Tissue React. 1995;17(5-6):211-7. PMID 8835632